CLINICAL TRIAL: NCT02579772
Title: Systemic Vascular Dysfunction in COPD Patients With Mild-to-moderate Airflow Obstruction: Pharmacological Treatment With N-acetylcysteine
Brief Title: Effects of N-acetylcysteine on Cardiorespiratory Control in COPD Patients With Mild-to-moderate Airflow Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. J. Alberto Neder, Principal Investigator, Queen's University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 6015083
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Results first posted 2018-06-14 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N-acetylcysteine (Active Comparator): Pharmacological treatment with N-acetylcysteine (NAC) pills
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): Treatment with placebo pills
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — Pharmacological treatment with N-acetylcysteine (NAC): 3 pills of 600 mg of NAC/day orally for 4 days prior to experimental procedures and 1 pill of 600 mg of NAC orally on the day of the experiment.
  Other Names: NAC pills
  Arms: N-acetylcysteine
Drug: Placebo — Placebo: 3 placebo pills/day orally for 4 days prior to experimental procedures and 1 placebo pill orally on the day of the experiment.
  Other Names: Placebo pills
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine whether pharmacological treatment with N-acetylcysteine improves central and peripheral cardiorespiratory control and physical capacity in COPD patients with mild-to-moderate airflow obstruction.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide. Cardiovascular complications constitute the main causes of poor physical capacity and healthcare resources utilization in COPD. There is emerging evidence that these impairments have a major impact on the health of patients with mild-to-moderate disease, the largest sub-population of COPD. This important problem, however, is currently neglected as no specific pharmacological treatment is offered to these patients. Recent studies indicate that vascular abnormalities are mediated, at least in part, by circulating inflammatory substances and direct damage of the arteries by oxygen radicals (oxidative stress). The current investigation will test the hypothesis that N-acetylcysteine (NAC), via its anti-inflammatory and antioxidant properties, improves systemic vascular function and physical capacity in COPD patients with mild-to-moderate airflow obstruction.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD with mild-to-moderate airflow obstruction as indicated by the low ratio between forced expiratory volume in one second and forced vital capacity (FEV1/FVC<0.7) together with post-bronchodilator FEV1≥60% predicted under optimized clinical treatment as judged by the accompanying physician

Exclusion Criteria:

* unable to perform all experimental procedures and/or provide informed consent;
* hospital admission in the previous 6 weeks;
* exercise training program in the previous 6 months;
* any condition that could interfere with the ability to exercise;
* diagnosed psychiatric or cognitive disorders;
* type I insulin-dependent diabetes mellitus;
* excessively over-weight (BMI>35kg/m²);
* other diagnosed cardiorespiratory disorders (e.g., chronic heart failure, peripheral artery disease).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Alberto Neder, MD, PhD, Principal Investigator — Queen's University

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- N-acetylcysteine, Then Placebo: Participants first received N-acetylcysteine (NAC; 3 pills of 600 mg of NAC/day orally for 4 days prior to experimental procedures and 1 pill of 600 mg of NAC orally on the day of the experiment). After a washout period of at least 7 days, they then received 3 placebo pills/day orally for 4 days prior to experimental procedures and 1 placebo pill orally on the day of the experiment.
- Placebo, Then N-acetylcysteine: Participants first received 3 placebo pills/day orally for 4 days prior to experimental procedures and 1 placebo pill orally on the day of the experiment. After a washout period of at least 7 days, they then received N-acetylcysteine (NAC; 3 pills of 600 mg of NAC/day orally for 4 days prior to experimental procedures and 1 pill of 600 mg of NAC orally on the day of the experiment).
Period: Overall Study
Arm/Group | N-acetylcysteine, Then Placebo | Placebo, Then N-acetylcysteine
Started | 8 | 5
Completed | 6 | 3
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Usage of additional antioxidants | 1 | 0
Not completed — flu-like illness, orthopedic trauma | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either N-acetylcysteine (NAC) or placebo pills
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Plasma Redox Status - Circulating Glutathione
Description: Fluorescent detection of plasma glutathione from samples collected during day 4 of each experimental arm (placebo vs. N-acetylcysteine)
Time Frame: pre-exercise value (day 4)
Measure: Mean (Standard Error); unit: micromolar
Groups:
- Placebo: 3 placebo pills/day orally for 4 days prior to experimental procedures and 1 placebo pill orally on the day of the experiment.
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
micromolar | 8.97 (0.61) | 7.05 (0.49)

2. Primary Outcome: Exercise Capacity - Time to Exhaustion
Description: Cycling time to exhaustion during day 4 of each experimental arm (placebo vs. N-acetylcysteine)
Time Frame: end-exercise value (Day 4)
Measure: Mean (Standard Error); unit: seconds
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
seconds | 336 (51) | 325 (47)

3. Secondary Outcome: Change in Central Cardiovascular Function - Cardiac Output
Description: During cycling to exhaustion during day 4 of each experimental arm (placebo vs. N-acetylcysteine)
Time Frame: end-exercise value (Day 4)
Measure: Mean (Standard Error); unit: liters/min
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
liters/min | 12.5 (1.0) | 12.1 (0.9)

4. Secondary Outcome: Change in Skeletal Muscle Deoxygenation - Dynamics (Mean Response Time)
Description: Mean response time (MRT) evaluated during cycling to exhaustion during day 4 of each experimental arm (placebo vs. N-acetylcysteine)
Time Frame: Day 4
Measure: Mean (Standard Error); unit: seconds
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
seconds | 19.0 (1.3) | 19.0 (2.5)

5. Secondary Outcome: Change in Skeletal Muscle Vascular Function - Capillary Blood Flow Dynamics (Mean Response Time)
Description: as for outcome 4
Time Frame: Day 4
Measure: Mean (Standard Error); unit: seconds
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
seconds | 65.4 (4.6) | 66.5 (7.6)

6. Secondary Outcome: Change in Pulmonary Oxygen Uptake - Dynamics (Mean Response Time)
Description: as for outcome 4
Time Frame: Day 4
Measure: Mean (Standard Error); unit: seconds
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
seconds | 63.0 (5.2) | 62.2 (4.4)

7. Secondary Outcome: Change in Pulmonary Ventilation - Minute Ventilation (VE)
Description: During cycling to exhaustion during day 4 of each experimental arm (placebo vs. N-acetylcysteine)
Time Frame: end-exercise value (Day 4)
Measure: Mean (Standard Error); unit: liters/min
Arm/Group | N-acetylcysteine | Placebo
Number analyzed (Participants) | 9 | 9
liters/min | 78.7 (7.6) | 75.8 (6.6)

ADVERSE EVENTS:
Time Frame: Adverse event data collected over the 4-day treatment period (NAC and placebo).
Arm/Group | N-acetylcysteine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N-acetylcysteine (N=9) | Placebo (N=9)
bloating, intestinal gas (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No